CLINICAL TRIAL: NCT01159288
Title: Phase II Trial of a Vaccination With Tumor Antigen-loaded Dendritic Cell-derived Exosomes on Patients With Unresectable Non Small Cell Lung Cancer Responding to Induction Chemotherapy
Brief Title: Trial of a Vaccination With Tumor Antigen-loaded Dendritic Cell-derived Exosomes
Acronym: CSET 1437
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IGR Dex2
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Advanced unresectable non small cell lung cancer; Responding or stabilized after induction chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

INTERVENTIONS:
Biological: Dex2 — * Metronomic dosage of Cyclophosphamide during 3 weeks (50mg/day orally) as reported 15, before specific treatment.
  * Induction immunotherapyIntradermal injections of Dex once a week during 4 consecutive weeks.(Peptides pulsed onto DC, sources of Dex: PRS pan-DR, MAGE-3 DP04, MAGE-1 A2, MAGE-3 A2, NY-ESO-1 A2 et MART-1 A2)
  * Continuation Immunotherapy: Intradermal injections of Dex every two weeks during 6 weeks.

SUMMARY:
Lung cancer is the worldwide leading cause of cancer death. In France, with 28,000 new cases per year, lung cancer is the 4th in terms of incidence but remains the leading cause of cancer death. The 5-year survival of lung cancer, all stages and all types, is very low, estimated at 12% among men and 16% among women in France. In advanced unresectable non small cell lung cancer, standard treatment relies on platinum-based induction chemotherapy. The median progression-free survival (PFS) in patients responding or stabilized after 4 chemotherapy cycles ranges from 2 to 2.8 months. Gustave Roussy and Curie institutes have developed an immunotherapy involving metronomic cyclophosphamide (mCTX) followed by vaccinations with tumor antigen-loaded dendritic cell-derived exosomes (Dex). mCTX inhibits Treg functions restoring T and NK cell effector functions and Dex are able to activate the innate and adaptive immunity. Phase I trials showed the safety and feasibility of Dex vaccines but no induction of T cells could be monitored in patients. Since 2007, we validated a new process for isolation of second generation Dex with improved immune stimulatory capacities. We propose a maintenance immunotherapy in 47 advanced unresectable NSCLC patients responding or stabilized after induction chemotherapy with Dex-based treatment to improve PFS rate at 4 months in these patients.

ELIGIBILITY:
Inclusion Criteria:

* advanced unresectable non small cell lung cancer
* responding or stabilizer after induction chemotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-05-19 (Actual); Primary Completion 2015-12-19 (Actual); Study Completion 2015-12-19 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Gustave Roussy, Villejuif, France